CLINICAL TRIAL: NCT06519877
Title: Modulation of the Gut Microbiome by Dietary Fiber to Improve Calcium Absorption and Bone Health in Older Men
Brief Title: Fiber and Calcium Absorption in Older Men
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: San Francisco VA Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: ENDB-009-23F; 24-41270 (Other: San Francisco VA Health Care System)
Record Dates: First submitted 2024-06-20; First posted 2024-07-25 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Aging

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into one of two groups at a 1:1 ratio in random permutated blocks of size 6. Each group will undergo 2 phases of intervention with soluble corn fiber 20g/day for 4 weeks and placebo (maltodextrin) for 4 weeks, with 4-weeks of washout in between. Group 1 will receive soluble corn fiber first followed by placebo, whereas group 2 will receive placebo first followed by soluble corn fiber. Outcomes will be assessed at the end of each intervention phase.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sachets of soluble corn fiber and placebo will be prepared and assigned randomization numbers by the investigational pharmacist at the San Francisco VA Health Care System. Participants, study staff, and those involved in outcome assessment will be blinded to the group assignment throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): Soluble corn fiber 20g/day x 4 weeks, washout period for 4 weeks, and placebo (maltodextrin) x 4 weeks.
  Interventions: Dietary Supplement: Soluble corn fiber
- Group 2 (Experimental): Placebo (maltodextrin) 20g/day x 4 weeks, washout period for 4 weeks, and soluble corn fiber x 4 weeks.
  Interventions: Dietary Supplement: Soluble corn fiber

INTERVENTIONS:
Dietary Supplement: Soluble corn fiber — Soluble corn fiber, also referred to resistant maltodextrin, is a type of dietary fiber made from corn starch. Soluble corn fiber is typically used to thicken processed foods and has been marketed as a prebiotic to improve digestive health.

SUMMARY:
Osteoporotic fractures are a major but underrecognized problem in men. There is growing evidence that low dietary fiber intake is a modifiable risk factor for age-related bone loss in men. Preclinical and human studies in adolescents and postmenopausal women suggest that dietary fiber intake influences bone metabolism by modulating the gut microbiome to augment intestinal calcium absorption, but it is unclear through what molecular mechanism and whether dietary fiber has the same effects in older men. In this crossover intervention study, the investigators will enroll and follow 30 older male Veterans to evaluate the effects of soluble corn fiber on intestinal calcium absorption and explore the contribution of the gut microbiome.

DETAILED DESCRIPTION:
Osteoporosis and associated fractures are a major problem in older men. One in four men over the age of 60 will sustain an osteoporotic fracture during his lifetime. Moreover, the mortality rate in men after fractures is nearly twice that in women. Despite the burden of fractures, little is understood about the pathogenesis of progressive bone loss in men. Studies point to dietary fiber as a potentially important mitigator of decline in bone mass, likely through increased intestinal calcium absorption and retention, as studied in adolescents, young men, and postmenopausal women. However, the effects of dietary fiber in older men have not been tested and the mechanism by which dietary fiber influences calcium absorption is unclear. The gut microbiome, which is crucial for host nutrient metabolism and hormone modulation, is a likely but underexplored mechanism.

The overall objective is to examine the effects of soluble corn fiber on intestinal calcium absorption with modulation of the gut microbiome in older men. The central hypothesis is that soluble corn fiber augments production of short-chain fatty acids by the gut microbiome, which modulates the production of systemic insulin-like growth factor 1 to increase calcium absorption and bone mass.

This study is a crossover intervention study on the effects of soluble corn fiber vs. placebo on intestinal calcium absorption and gut microbiome composition and function in 30 older male Veterans 60 years of age. Participants will be randomized 1:1 to sequential soluble corn fiber 20g/day vs. placebo for4 weeks each with a 4-week washout period. Individualized doses of calcium and vitamin D supplementation will also be provided through out the study period. Study measurements at the end of each intervention include intestinal calcium absorption via a dual stable isotope method, detailed gut microbiome characterization with metagenomics and metabolomics, dietary assessment, calciotropic hormones, and bone turnover marker levels. Baseline bone density and microstructure will also be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Male Veterans 60 years of age

Exclusion Criteria:

* History of malabsorption
* Hypercalcemia (corrected Ca > 10.2 mg/dL)
* Vitamin D insufficiency (25OHD < 30 ng/mL)
* Chronic kidney disease stage 3B or worse (CrCl < 45 mL/min)
* Severe hypogonadism (AM fasting serum total testosterone < 150 ng/dL)
* Daily use of proton pump inhibitor
* Use of medication(s) known to affect calcium metabolism
* Use of medications or supplements that could impact gut microbiota in the previous 3 months (antibiotics or commercially available probiotics or prebiotics.
* Presence of a condition or abnormality that in the opinion of the Investigator that would compromise the safety of the patient or the quality of the data.

Min Age: 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Intestinal fractional calcium absorption | At week 4 and week 12 of study participation (at the end of each treatment phase x2)
  Dual stable calcium isotopic tracer method

SECONDARY OUTCOMES:
Biochemical markers of bone turnover | At week 4 and week 12 of study participation (at the end of each treatment phase x2)
  Blood draw
Calciotropic hormones | At week 4 and week 12 of study participation (at the end of each treatment phase x2)
  Blood draw
Gut microbial profiling | At week 4 and week 12 of study participation (at the end of each treatment phase x2)
  Stool collection
Adherence, tolerability, and acceptability | Throughout study period, an average of 12 weeks
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Karin C Wu, MD, Principal Investigator — San Francisco VA Medical Center, San Francisco, CA
Locations (1):
- San Francisco VA Medical Center, San Francisco, CA, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No